CLINICAL TRIAL: NCT02053532
Title: Functional Brain Imaging in PTSD
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S13-00313
Record Dates: First submitted 2014-01-22; First posted 2014-02-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Trauma
Keywords: Trauma; Post-traumatic stress disorder (PTSD); Imaging; Neuroimaging; F-18-fluorodeoxyglucose (FDG)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Positron emission tomography/magnetic resonance imaging
  Interventions: Procedure: Positron emission tomography/magnetic resonance imaging

INTERVENTIONS:
Procedure: Positron emission tomography/magnetic resonance imaging — Positron emission tomography/magnetic resonance (PET/MR) imaging using 18-F-fluorodeoxyglucose (FDG) as radio tracer
  Other Names: PET Imaging

SUMMARY:
Patients with post-traumatic stress disorder (PTSD) have abnormalities in the function of the amygdala and medial prefrontal cortex (particularly anterior cingulate), in addition to abnormalities of hippocampal volume. In this pilot study we propose to use the combined positron emission tomography/magnetic resonance (PET/MR) scanner and F-18-fluorodeoxyglucose (FDG, an analog of glucose, the most commonly used PET ligand) to examine brain function and directly correlate the data with the intrinsic functional connectivity of brain circuits that are responsible for social, emotional and cognitive processing in both individuals with PTSD and group-matched trauma controls (TC) and healthy controls (HC). Once the machine is validated, we will then use a more specific biomarker to better understand the neurochemical factors that contribute to individual differences in PTSD. Thus, the data obtained from this pilot study will guide our future molecular imaging studies. The link between general brain function, specific molecular target and the intrinsic functional connectivity of brain circuits that are responsible for social, emotional and cognitive processing in PTSD, TC and HC will be explored.

ELIGIBILITY:
For Patients with post-traumatic stress disorder (PTSD)

Inclusion criteria:

1. Age 18-55 years old
2. Currently diagnosed with PTSD and symptomatic with a Clinician-Administered PTSD Scale (CAPS) score > 50

Exclusion criteria:

1. any primary Axis I disorder other than PTSD (e.g. psychosis)
2. medical or neurological illnesses likely to affect physiology or anatomy, i.e. uncontrolled hypertension, cardiovascular disorders
3. a history of drug (including benzodiazepines (BZD)) dependence (Diagnostic and Statistical Manual (DSM) IV criteria) within 1 year of the study and lasting longer than 2 years, except for alcohol dependence
4. current pregnancy (as documented by pregnancy testing at screening or on the day of PET imaging study)
5. current breast feeding
6. nicotine dependence
7. suicidal ideation or behavior
8. general magnetic resonance imaging (MRI) exclusion criteria, i.e. pacemakers, metals in the body;
9. Human immunodeficiency virus (HIV) (due to possible neuropsychiatric effects)
10. Hepatitis B or C (due to possible neuropsychiatric effects)
11. use of opioid medications within 2 weeks of the positron emission tomography (PET) study
12. having an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participation in the study
13. seriously claustrophobic
14. blood donation within 8 weeks prior to the study
15. positive alcohol breathalyzer test
16. Abnormal thyroid test indicated by thyroid stimulating hormone (TSH) < .15 mlU/L and/or thyroxine (T4) > 18 mcg/dL
17. Glucose > 200 mg/dL on two separate days

For Healthy Subjects

Inclusion criteria:

1. Age 18-55 years old
2. No personal or first-degree family history of any Axis I diagnosis

Exclusion criteria:

1. . any history or current primary Axis I disorder ;
2. . medical or neurological illnesses likely to affect physiology or anatomy, i.e. uncontrolled hypertension, cardiovascular disorders;
3. . a history of drug (including benzodiazepines [BZD]) dependence (DSM IV criteria) within 1 year of the study and lasting longer than 2 years, except for alcohol dependence;
4. . current pregnancy (as documented by pregnancy testing at screening or on the day of PET imaging study);
5. . current breast feeding;
6. . nicotine dependence;
7. . suicidal ideation or behavior;
8. . general MRI exclusion criteria, i.e. pacemakers, metals in the body;
9. . HIV (due to possible neuropsychiatric effects);
10. . Hepatitis B or C (due to possible neuropsychiatric effects);
11. . use of opioid medications within 2 weeks of the PET study;
12. . having an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participation in the study;
13. . seriously claustrophobic;
14. . blood donation within 8 weeks prior to the study;
15. . positive alcohol breathalyzer test;
16. . Abnormal thyroid test indicated by TSH < .15 mlU/L and/or T4 > 18 mcg/dL;
17. . Glucose > 200 mg/dL on two separate days;
18. . Does not have a lifetime history of trauma.

For Healthy Subjects with Trauma ("Trauma Controls")

Inclusion criteria:

1. . Age 18-55 years old;
2. . No personal or first-degree family history of any Axis I diagnosis;
3. . Has a lifetime history of trauma.

Exclusion criteria:

1. . any history or current primary Axis I disorder ;
2. . medical or neurological illnesses likely to affect physiology or anatomy, i.e. uncontrolled hypertension, cardiovascular disorders;
3. . a history of drug (including benzodiazepines [BZD]) dependence (DSM IV criteria) within 1 year of the study and lasting longer than 2 years, except for alcohol dependence;
4. . current pregnancy (as documented by pregnancy testing at screening or on the day of PET imaging study);
5. . current breast feeding;
6. . nicotine dependence;
7. . suicidal ideation or behavior;
8. . general MRI exclusion criteria, i.e. pacemakers, metals in the body;
9. . HIV (due to possible neuropsychiatric effects);
10. . Hepatitis B or C (due to possible neuropsychiatric effects);
11. . use of opioid medications within 2 weeks of the PET study;
12. . having an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participation in the study;
13. . seriously claustrophobic;
14. . blood donation within 8 weeks prior to the study;
15. . positive alcohol breathalyzer test;
16. . Abnormal thyroid test indicated by TSH < .15 mlU/L and/or T4 > 18 mcg/dL;
17. . Glucose > 200 mg/dL on two separate days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are between the age range of 18 to 65, are medically healthy and currently not taking any medications to treat any medical illness, and either have no history of post-traumatic stress disorder (PTSD) or have been diagnosed with PTSD.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
F-18- fluorodeoxyglucose (FDG) metabolism in the brain of healthy controls (HC) vs trauma controls (TC) vs individuals with post-traumatic stress disorder (PTSD) | Two months
  In this pilot study we propose to use the combined positron emission tomography/magnetic resonance (PET/MR) scanner and F-18-fluorodeoxyglucose (FDG, an analog of glucose, the most commonly used PET ligand) to examine brain function and directly correlate the data with the intrinsic functional connectivity of brain circuits that are responsible for social, emotional and cognitive processing in both individuals with post-traumatic stress disorder (PTSD) and group-matched trauma controls (TC) and healthy controls (HC). These groups are matched based on gender, age and ethnicity. Once the machine is validated, we will then use a more specific biomarker to better understand the neurochemical factors that contribute to individual differences in PTSD. The link between general brain function, specific molecular target and the intrinsic functional connectivity of brain circuits that are responsible for social, emotional and cognitive processing in PTSD, TC and HC will be explored.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU School of Medicine, New York, New York, United States